CLINICAL TRIAL: NCT00003607
Title: Phase III Randomized Study of Radiotherapy to the Prostate With or Without Radiotherapy to the Pelvis in Patients With Stage I, II, or III Adenocarcinoma of the Prostate
Brief Title: Radiation Therapy in Treating Patients With Stage I, Stage II, or Stage III Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066684; FRE-FNCLCC-GETUG-01; EU-98029
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known whether radiation therapy to the prostate and pelvis is more effective than radiation therapy to the prostate alone in treating prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy to the prostate with or without radiation to the pelvis in treating patients with stage I, stage II, or stage III prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the survival without recurrence and overall survival of patients with stage I, II, or III adenocarcinoma of the prostate after receiving radiotherapy to the prostate with or without radiotherapy to the pelvis.
* Compare the toxic effects of these two regimens in these patients.
* Compare the quality of life of patients treated with these regimens.
* Determine the prognostic factors of progression in these patients.
* Analyze the site of relapse (prostate, pelvic lymph nodes, metastases) in case of progression in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by participating center and prognostic group (poor vs good prognosis).

Patients are randomized to one of two treatment arms.

* Arm I: Patients receive pelvic irradiation plus local prostate irradiation.
* Arm II: Patients receive local prostate irradiation only. Radiotherapy in both arms is administered 5 days a week for 7 weeks.

Quality of life is assessed before therapy, 12 months after therapy, and then annually thereafter.

Patients are followed at 2 and 6 months and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 450 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven adenocarcinoma of the prostate

  * Stage I (T1b or T1c, N0, M0)
  * Stage II (T2, N0, M0)
  * Stage III (T3, N0, M0)
* Poor prognosis (high risk of lymph node invasion) defined as meeting at least 1 of the following criteria:

  * Gleason score at least 7
  * Prostate-specific antigen (PSA) at least 3 times upper limit of normal (ULN)
  * T3 OR
* Good prognosis defined as meeting 1 of the following criteria:

  * T1b or T2
  * T1c with Gleason score less than 7 and PSA less than 3 times ULN
* No metastases by bone scans or chest x-ray

PATIENT CHARACTERISTICS:

Age:

* 75 and under

Performance status:

* Karnofsky 70-100%

Life expectancy:

* More than 10 years

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other malignancy within the past 10 years except basal cell skin cancer
* No adenopathies

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* At least 2-6 months since prior hormonal therapy, if duration no greater than 4-8 months
* No concurrent luteinizing hormone-releasing hormone agonists
* No concurrent anti-androgen therapy
* No concurrent hormonal therapy in high-risk group

Radiotherapy:

* No prior pelvic radiotherapy

Surgery:

* No prior lymphadenectomy
* No prior surgical castration
* No prior prostatectomy
* At least 1 month since prior transurethral resection

Max Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 1997-12; Primary Completion 2002-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Pommier, MD, Study Chair — Centre Leon Berard
Locations (23):
- France (23):
  - Centre Paul Papin, Angers
  - Centre Hospitalier d'Annecy, Annecy
  - Institut Bergonie, Bordeaux
  - Centre Regional Francois Baclesse, Caen
  - Centre de Radiotherapie du Parc, Chalon-sur-Saône
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Centre Oscar Lambret, Lille
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Clinique de la Sauvegarde - Clinique Jeanne D'Arc, Lyon
  - Clinique de la Sauvegarde, Lyon
  - Centre Leon Berard, Lyon
  - Institut J. Paoli and I. Calmettes, Marseille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Hopital d'Instruction des Armees du Val de Grace, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - CHG Roanne, Roanne
  - Clinique de l'Orangerie, Strasbourg
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Centre Marie Curie, Valance

REFERENCES:
- [Result] Pommier P, Chabaud S, Lagrange JL, Richaud P, Lesaunier F, Le Prise E, Wagner JP, Hay MH, Beckendorf V, Suchaud JP, Pabot du Chatelard PM, Bernier V, Voirin N, Perol D, Carrie C. Is there a role for pelvic irradiation in localized prostate adenocarcinoma? Preliminary results of GETUG-01. J Clin Oncol. 2007 Dec 1;25(34):5366-73. doi: 10.1200/JCO.2006.10.5171. PMID 18048817
- [Result] Pommier P, Perol D, Lagrange J, et al.: Does pelvis and prostate radiation therapy compared to prostate radiation therapy alone improve survival in patients with non metastatic prostate carcinoma? Preliminary results of the prospective randomized GETUG 01 trial. [Abstract] Int J Radiat Oncol Biol Phys 63 (Suppl 1): A-33, S19, 2005.